CLINICAL TRIAL: NCT00751140
Title: Merits of Performing a Modified Template Retroperitoneal Lymph Node Dissection at Time of Nephroureterectomy for Urothelial Carcinoma of the Upper Urinary Tract
Brief Title: Merits of Performing a Modified Template Retroperitoneal Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-15441; 10718 (Other: USF IRB)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2012-12

CONDITIONS: Cancer of the Urinary Tract
Keywords: surgical candidates; upper urinary tract; urothelial carcinoma; lymph node dissection
MeSH Terms: conditions — Urologic Neoplasms; Carcinoma, Transitional Cell | interventions — Lymph Node Excision; Nephroureterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymph Node Dissection at Time of Nephroureterectomy (Experimental): A prospective single-arm two-stage phase II study to allow for analysis of the treatment-specific outcomes and disease-specific survival of patients treated with open or laparoscopic nephroureterectomy and bladder cuff excision along with a lymph node dissection (modified template retroperitoneal lymph node dissection).
  Interventions: Procedure: Lymph Node Dissection

INTERVENTIONS:
Procedure: Lymph Node Dissection — The lymph nodes will be sent to pathology for review.
  Other Names: nephroureterectomy

SUMMARY:
The primary objective is to show that performing a lymph node dissection may detect occult nodal metastasis in this patient population whereby providing important diagnostic information, with potential therapeutic benefits in patients with isolated nodal metastases.

In case of urothelial carcinoma of the upper urinary tract (a cancer originating from the inner lining of the urinary tract) requiring the removal of the kidney, ureter, and cuff of bladder (a surgical termed a nephroureterectomy). Previous studies in urothelial carcinoma of the bladder, have shown that doing a lymph node dissection (surgically removing the lymph nodes) may improve survival, or at least give an idea of what patients may need chemotherapy (drugs to control the cancer cells that are outside the kidney-ureter) earlier (before the nodes are enlarged in the imaging studies).

DETAILED DESCRIPTION:
Participants will have a nephroureterectomy (taking the kidney and the ureter). Investigators will also be doing a lymph node dissection (taking the patient's lymph nodes in the same side of the kidney) to look for malignancy outside of the kidney and ureter. The lymph nodes will be sent to pathology for review.

Study visits will be scheduled 10 to 14 days after surgery for removal of stitches and analysis of the patient's pathology report.

The following procedures will be done:

* History and physical examination, urinary cytology (test to look for malignant cells in the urine) and surveillance cystoscopy (procedure to look inside the urethra and bladder which is performed in the office under local anesthesia) every 3 months for the first 2 years after treatment, every 6 months for the next 2 years and yearly thereafter if the patient is free from recurrence.
* Radiographic studies including chest x-ray and abdomino-pelvic computed tomography (CAT scans) will be performed every 6 months for the first 2 years and then yearly thereafter.
* Bone scan (special imaging study to look for cancer spread in bone) in case of bone pain or elevated alkaline phosphatase level.

After surgery patients will be followed every 3 months for the first 2 years after treatment, every 6 months for the next 2 years and yearly thereafter if they are free from recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected transitional cell carcinoma of the upper urinary tract which are deemed surgical candidates
* Negative visible retroperitoneal or peri-hilar lymphadenopathy on pre-operative radiographic studies. Defined as the absence of suspicious abdominal, retroperitoneal, or pelvic lymphadenopathy (defined as > 1 centimeter [cm]) on pre-operative radiographic imaging (Abdominal and pelvic computed tomography [CT] or magnetic resonance imaging [MRI] if CT contraindicated). Imaging studies can be done at Moffitt or at a local facility of the patient's choice. All imaging studies are going to be reviewed at Moffitt.
* Note: Nodal involvement will depend on the size of the lymph node enlargement; usually nodes of more than 2 cm are associated with malignancy. With a threshold of 1cm, false negative rates for microscopic metastases are low (4%) and false positive rates are between 3 to 43% according to the literature. Because the aim of the study will be to perform a lymph node dissection in patients with non-metastatic disease based on pre-operative evaluation, 1 cm will be the threshold used. Nodes of more than 1 cm will be considered positive and those patients will be excluded as is mentioned in the protocol. Biopsy will not be included as part of the protocol as those potential patients with nodes of more than 1 cm will be excluded.
* No other suspected sites of metastasis on pre-operative radiographic imaging

Exclusion Criteria:

* Patients with visible lymph node metastasis on pre-operative radiographic studies. Defined as >1cm abdominal, retroperitoneal or pelvic lymphadenopathy
* Patients with suspected sites of distant metastasis on pre-operative imaging. (Patients with suspected bony metastases will require a bone scan.)
* Patients with suspected transitional cell carcinoma of the upper urinary tract with significant comorbidities making them non-surgical candidates
* Patients with non-transitional cell carcinoma of the upper urinary tract will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Spiess, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Prospective clinical trial of the feasibility and safety of modified retroperitoneal lymph node dissection at time of nephroureterectomy for upper tract urothelial carcinoma. — https://www.ncbi.nlm.nih.gov/pubmed/22564727
- See also: Prospective clinical trial of the feasibility and safety of modified retroperitoneal lymph node dissection at time of nephroureterectomy for upper tract urothelial carcinoma — http://onlinelibrary.wiley.com/doi/10.1111/j.1464-410X.2012.11170.x/full

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sample: Up to 30 patients with a diagnosis of urothelial carcinoma of the upper urinary tract in the absence of pre-operative (radiographic) lymphadenopathy or other areas of suspected metastatic disease were planned to serve as the investigators' study sample population.
Groups:
- Lymph Node Dissection at Time of Nephroureterectomy: A prospective single-arm two-stage phase II study to allow for analysis of the treatment-specific outcomes and disease-specific survival of patients treated with open or laparoscopic nephroureterectomy and bladder cuff excision along with a lymph node dissection (modified template retroperitoneal lymph node dissection).
  Lymph Node Dissection : The lymph nodes will be sent to pathology for review.
Period: Overall Study
Arm/Group | Lymph Node Dissection at Time of Nephroureterectomy
Started | 20
Completed | 19
Not Completed | 1
Not completed — benign angioma excluded from analysis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lymph Node Dissection at Time of Nephroureterectomy
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 69 [42 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologically Proven Lymph Node Metastasis
Description: The number of participants having pathologically proven lymph node metastasis at the time of radical nephroureterectomy (RNU) and modified retroperitoneal lymph node dissection (RPLND).
  The primary endpoint is the detection via lymph node dissection of pathological node positive urothelial carcinoma in patients treated with open or laparoscopic nephroureterectomy for upper tract urothelial cancer.
Time Frame: Up to 4 years
Population: All evaluable participants. On histopathological review, one patient had a benign angioma and was excluded from the final data analysis.
Measure: Number; unit: participants
Arm/Group | Lymph Node Dissection at Time of Nephroureterectomy
Number analyzed (Participants) | 19
participants | 1

2. Secondary Outcome: Surgical Outcomes: Mean Lymph Node Count
Description: The mean (range) total lymph node count and lymph node count per procedure category. Between 2009 and 2011, patients with suspected upper urinary tract urothelial carcinoma (UUT-UC) underwent open, laparoscopic, or robot-assisted radical nephroureterectomy (RNU) with modified retroperitoneal lymph node dissection (RPLND).
Time Frame: 2 years
Population: Total Participants and Participants Per Procedure Category
Measure: Mean (Full Range); unit: Lymph Nodes
Groups:
- Total Lymph Node Count: Total Lymph Node Count for All Participants
- Open RNU Lymph Node Count: Lymph Node Count for Open RNU Procedure Group
- Laparoscopic RNU Lymph Node Count: Lymph Node Count for Laparoscopic RNU Procedure Group
- Robot-assisted RNU Lymph Node Count: Lymph Node Count for Robot-assisted RNU Procedure Group
Arm/Group | Total Lymph Node Count | Open RNU Lymph Node Count | Laparoscopic RNU Lymph Node Count | Robot-assisted RNU Lymph Node Count
Number analyzed (Participants) | 20 | 9 | 4 | 7
Lymph Nodes | 7 [2 to 17] | 7 [2 to 17] | 8 [3 to 14] | 6 [2 to 10]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lymph Node Dissection at Time of Nephroureterectomy
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymph Node Dissection at Time of Nephroureterectomy (N=19)
Chylous leak requiring surgical exploration - Grade IIIb (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymph Node Dissection at Time of Nephroureterectomy (N=19)
Blood Transfusion - Grade II (Renal and urinary disorders) | 6 (6)
Postoperative ileus - Grade II (Renal and urinary disorders) | 1 (1)
Chylous leak managed conservatively - Grade II (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size was small because it was a single institution study. It was thus underpowered to achieve a cancer-specific endpoint pertaining to the oncological merit of performing a modified RPLND in the context of UUT-UC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes